CLINICAL TRIAL: NCT02478580
Title: The Effects of Armodafinil (Nuvigil) on Postoperative Recovery of OSA (Obstructive Sleep Apnea) and Obese Patients
Brief Title: Armodafinil (Nuvigil), Postoperative Recovery of OSA (Obstructive Sleep Apnea) and Obese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Enas Kandil, Medical Doctor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10-041
Record Dates: First submitted 2015-06-08; First posted 2015-06-23 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Obesity; Premature Recovery From Anesthesia
Keywords: Obstructive Sleep Apnea; Anesthesia Recovery Period
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nuvigil (Experimental): A single oral dose of Nuvigil at 150mg dose in preoperative area
  Interventions: Drug: Nuvigil
- Placebo (Placebo Comparator): A single oral placebo will be given in preoperative area
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nuvigil — Patients will receive Nuvigil before the surgery
  Other Names: Armodafinil
  Arms: Nuvigil
Drug: Placebo — Placebo will be given before surgery
  Other Names: Oral placebo
  Arms: Placebo

SUMMARY:
Obstructive sleep apnea (OSA) and obesity is associated with increased perioperative morbidity and mortality. This group of patients is at risk of perioperative desaturations which can be worsened by perioperative sedatives and narcotics needed for surgery. OSA patients might also need to spend the night in intensive care for more frequent monitoring for any desaturations episodes especially if the patient will be requiring multiple intravenous narcotic boluses for pain control. Several studies have looked into the most appropriate way to manage these patients and some recommendations have been made to avoid outpatient surgery with close monitoring for first 24 hours after surgery specifically if patient will require intravenous postoperative narcotics.

Nuvigil (Armodafinil) is a wake promoting agent (Cephalon inc., West Chester, PA) that's FDA approved for excessive daytime sleepiness in narcolepsy, shift work sleep disorder, and obstructive sleep apnea. The precise mechanism(s) through which armodafinil (R-enantiomer) or modafinil (mixture of R- and S-enantiomers) promote wakefulness is unknown.

Nuvigil is longer acting product which is similar in action to Modafinil however is much cheaper. Nuvigil has not been previously studied for postoperative recovery. The investigators intend to study the effects of Nuvigil on postoperative recovery time and wakefulness in obstructive sleep apnea and obese patients.

DETAILED DESCRIPTION:
Modafinil has been shown to improve recovery after general anesthesia in a small pilot study which involved 30 patients. In these study, patients were given one dose of Modafinil 200mg po versus placebo after surgery when patient tolerating po with a sip of water and were discharged home. They were asked to assess their fatigue, alertness and energy level during the following 24 hrs. Modafinil was found to significantly reduce fatigue and improves feelings of alertness and energy in postoperative patients. It was concluded that patients recovering from general anesthesia can significantly benefit from Modafinil.

A more recent study looked at the perioperative use of Modafinil in 67 patients presenting for lithotripsy requiring sedation. Goal was to asses improvement in recovery compared to placebo. Patients were randomized to 4 groups 1 and 2 received midazolam/ fentanyl sedation plus Modafinil 200mg po given 1 hr before sedation versus placebo, the other two received remifentanil / propofol infusion plus Modafinil 20 mg po versus placebo. Groups were compared using the digital symbol substitution test (DSST), trail making test (TMT), observer scale of sedation and analgesia (OAA/S) and Aldrete score and they found no statistical significant difference between groups. However they measured the Verbal rating scale (VRS) scores for secondary outcome variables e.g. energy, tiredness and dizziness were also recorded before and after treatment. They concluded that Modafinil reduces patient-reported tiredness after sedation/analgesia however does not improve recovery in terms of objective measures of patient psychomotor skills.

Nuvigil is longer acting product which is similar in action to Modafinil and has not been previously studied for postoperative recovery. We intend to study the effects of Nuvigil on postoperative recovery time and wakefulness in obstructive sleep apnea patients and obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient presented for surgery under general anesthesia
* Documented OSA
* Patients with BMI above 35

Exclusion Criteria:

* Coronary Artery Disease or Myocardial infarcts
* Mitral valve prolapse
* Cyclosporine, contraceptive drugs
* Known allergic reaction to Modafinil or any of its products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enas Kandil, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nuvigil: A single oral dose of Nuvigil 150mg in preoperative area
  NUVIGIL: Patient will receive Nuvigil before the surgery
- Control: Placebo in preoperative area
  Patient will receive placebo before the surgery
Period: Overall Study
Arm/Group | Nuvigil | Control
Started | 34 | 33
Completed | 34 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patient with obstructive sleep apnea undergoing surgery
Groups:
- Control: Placebo in preoperative area
- Total: Total of all reporting groups
Arm/Group | Nuvigil | Control | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (12.7) | 54.7 (10.8) | 53.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 29 | 29 | 58
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Care Unit (PACU) Recovery Time
Description: Participants will be followed for the duration of PACU stay, an expected average of 3 hours.
Time Frame: Immediate postoperative period (up to 3 hours)
Population: Patient with obstructive sleep apnea undergoing surgery
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Nuvigil | Control
Number analyzed (Participants) | 34 | 33
Minutes | 98.2 (58.2) | 95 (60.7)

2. Secondary Outcome: The Aldrete Score
Description: Aldrete score used for readiness of PACU discharge by assigning numeric values to the criteria including activity, respiration, circulation, consciousness, and color. Each criterion is rated from 0 to 2, with a maximum score of 10. Scores in the range of 9 to 10 are considered satisfactory for PACU discharge.
Time Frame: 2 hours after extubation
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: A single oral placebo will be given in preoperative area
  Nuvigil: Patients will receive Nuvigil before the surgery
Arm/Group | Nuvigil | Placebo
Number analyzed (Participants) | 34 | 33
units on a scale | 9.4 (0.27) | 9.3 (0.26)

ADVERSE EVENTS:
Time Frame: Postoperative 24-h period.
Description: Fatigue was assessed during postoperative 24-h period.
Groups:
- Nuvigil: A single oral dose of Nuvigil 150 mg in preoperative area
  NUVIGIL: Patient will receive Nuvigil before the surgery
Arm/Group | Nuvigil | Control
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No